CLINICAL TRIAL: NCT03618758
Title: Safety and Efficacy of Intraperitoneal Paclitaxel in Gastric Cancer Patients With Peritoneal Metastasis Receiving Systemic Chemotherapy
Brief Title: Intraperitoneal Paclitaxel Plus Systemic mFOLFOX6
Acronym: IPLUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry); B. Braun Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH_GS_IPEC
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer Stage IV; Peritoneal Carcinomatosis; Intraperitoneal Paclitaxel; mFOLFOX6
Keywords: Gastric cancer; Peritoneal carcinomatosis; Intraperitoneal chemotherapy; Paclitaxel; FOLFOX
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Paclitaxel; genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gastric Cancer with Peritoneal Carcinomatosis (Experimental): Intraperitoneal Chemotherapy (Paclitaxel) + Systemic mFOLFOX6(5-FU, Oxaliplatin, Leucovorin)
  Interventions: Drug: Paclitaxel; Drug: mFOLFOX6 regimen

INTERVENTIONS:
Drug: Paclitaxel — Intraperitoneal application of Paclitaxel Phase 1: Dose determination of Paclitaxel (Recommended Dose) Starting from 40mg/m² upto 100mg/m² maximum
  Phase 2: Intraperitoneal Paclitaxel with recommended dose
  Other Names: (Genexol®)
Drug: mFOLFOX6 regimen — Systemic mFOLFOX6: 5-FU(2400mg/m²), Oxaliplatin(100mg/m²), Leucovorin(100mg/m²)

SUMMARY:
Treatment for stage 4 gastric cancer with peritoneal carcinomatosis has been unchanged for decades. The median survival for stage 4 gastric cancer is 9-14 months with systemic chemotherapy. Intraperitoneal chemotherapy in combination with systemic chemotherapy is under many clinical trials mainly in Japan, and are showing promising results.

This is Korea's first clinical trial on Intraperitoneal Paclitaxel with Systemic mFOLFOX6 chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of gastric origin, primary or recurrent
* Identification of Peritoneal seeding by CT or diagnostic laparoscopy
* Patients confirmed to receive mFOLFOX6 on multidisciplinary outpatient clinic
* No previous history of chemotherapy or 4week after the last chemotherapy for gastric cancer
* Labs adequate for chemotherapy (within 2 weeks of enrollment)
* Absolute Neutrophil Count: ≧ 1,500/mm³
* Hemoglobin level: ≧ 8.0g/dL
* Platelet Count: ≧ 10×104/mm³
* AST (GOT), ALT (GPT): ≦ 100U/L
* Total Bilirubin: ≦ 2.0mg/dL
* Creatinine Clearance (CCl): ≧ 50mL/min
* ECOG 0 - 2
* Her-2 negative on endoscopic biopsy
* Age ≧ 20, < 80
* Signed Informed consent form

Exclusion Criteria:

* Patients with other major medical disease or malignant tumors other than gastric cancer
* Contraindication to 5-FU, Oxaliplatin, Leukovorin or Paclitaxel
* Pregnant, breast-feeding women or with birth plan
* Patients refusing treatment

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Dose determination (Phase 1) | 1 Year
  Dosage determination of Intraperitoneal Paclitaxel
Overall survival (Phase 2) | 1 Year
  1 year Overall survival with determined dose from Phase 1

SECONDARY OUTCOMES:
Progression-free survival | 1 Year
  1 year Progression-free survival
Toxicity ratio | 3 Years
  Toxicity occurrence ratio by CTCAE V.4
Tumor response | 3 Years
  Tumor response with RECIST criteria V.1.1 and Peritoneal Regression Grading Score(PRGS) system
Conversion surgery ratio | 3 Years
  Conversion surgery after stable disease or regression

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Ho Kim, M.D., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided